CLINICAL TRIAL: NCT00186667
Title: An Open Label Study of Sirolimus as Primary Therapy for the Treatment of Chronic GVHD Following Allogeneic Bone Marrow Transplant
Brief Title: Sirolimus as Primary Therapy for the Treatment of Chronic Graft Versus Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-SQL 75568; BMT81 (Other: OnCore)
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Graft vs Host Disease; Blood and Marrow Transplant (BMT)
MeSH Terms: conditions — Graft vs Host Disease | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Procedure: high dose chemotherapy and autologous hematopoietic cell transplant

SUMMARY:
Evaluate the clinical activity of sirolimus in combination with cyclosporine and corticosteroids as first line therapy for the treatment of chronic Graft Versus Host Disease.

DETAILED DESCRIPTION:
An Open Label Study of Sirolimus as Primary Therapy for the Treatment of Chronic GVHD Following Allogeneic Bone Marrow Transplant

ELIGIBILITY:
Inclusion Criteria:- active chronic GvHD

* ANC > 1000/mm^3
* therapeutic cyclosporine Exclusion Criteria:- uncontrolled systemic infection
* elevated serum creatinine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1999-01; Primary Completion 2000-01 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of clinical activity of sirolimus in combination with cyclosporine and corticosteroids as first line therapy for the treatment of chronic Graft Versus Host Disease.

SECONDARY OUTCOMES:
Evaluate the safety of clinical activity of sirolimus in combination with cyclosporine and corticosteroids as first line therapy for the treatment of chronic Graft Versus Host Disease.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Johnston, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States